CLINICAL TRIAL: NCT04648904
Title: Fractionation Accelerated Beyond Standard Therapy for Post-Mastectomy Radiotherapy in Patients With Reconstructions (FAST-R Trial): A Prospective Non-inferiority Trial of Ultra-compressed Treatment
Brief Title: Study of a Shortened Radiation Therapy Schedule in People With Breast Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-513
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Invasive Breast Cancer; Post-mastectomy
Keywords: AJCC Stage IIa - IIIa; Pathologic stage T0N1a-2a; Pathologic stage T1N1a-2a; Pathologic stage T2N1a-2a; Pathologic stage T3N0-2a, all M0 status; Radiotherapy; Ultra-compressed Treatment; 20-513; T3N0 patients
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: This is a single-arm, single-site, prospective non-inferiority trial of PMRT delivered in the compressed FAST FORWARD schedule.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-Mastectomy Radiotherapy (Experimental): Treatment will consist of PMRT delivered using external beam RT techniques to a dose of 26 Gy in 5 fractions of 5.2 Gy delivered on consecutive weekdays with an optional chest wall boost of 5.2 Gy for 1-2 fractions or an alternate boost schedule of 2.5 Gy for 1-4 fractions at the discretion of the treating physician.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — A total dose of 26 Gy in 5 fractions will be given once daily over 5 consecutive weekdays (or within 10 consecutive weekday to allow for treatment delays, interruptions, logistical problems, scheduling issues and weekends/holidays).

SUMMARY:
The purpose of this study is to see whether providing radiation on a shortened (compressed) schedule of 5 days in a row is a safe and effective approach to prevent cancer from coming back in people who have had a mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients with invasive breast cancer who have had mastectomy and have a chest wall reconstruction in progress or completed.
* Age ≥ 30 years
* Final AJCC Stage IIa - IIIa (pathologic stage T0N1a-2a, T1N1a-2a, T2N1a-2a, T3N0-2a, all M0 status). Pathological stage for all patients not receiving neoadjuvant chemotherapy. Higher of the clinical or pathological T and N stage, if receiving neoadjuvant chemotherapy. T3N0 patients, either clinically by imaging before neoadjuvant chemotherapy, or by pathological stage at the time of surgery, are eligible. Exceptions to these criteria (e.g. for T4 or N3 patients) are possible after discussion with PI.
* Histologically negative tumor margin.
* ECOG Performance Status of 0 or 1

Exclusion Criteria:

* Patients with distant metastasis.
* Patients who are pregnant or breastfeeding.
* Prior radiation therapy to the ipsilateral or contralateral breast or thorax.
* All patients with clinical, radiographic or pathological T4, N3 or involved internal mammary disease (N1b, N1c, and N2b) will not be eligible to enroll.
* Medical condition such as uncontrolled infection (including HIV), uncontrolled diabetes mellitus, or connective tissue diseases (lupus, systemic sclerosis, or other collagen vascular diseases) that, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have "currently active" malignancies if they have completed therapy and are considered by their physicians to be at <5% risk of relapse within 3 years.
* Concomitant anti-neoplastic treatment is not allowed during protocol treatment and should be completed at least 2 weeks prior to commencement of protocol treatment, with resolution of associated acute toxicities. However endocrine therapies (tamoxifen or aromatase inhibitors), anti-HER2 therapy and bisphosphonates are permitted without restriction even during protocol treatment. Standard-of-care maintenance treatments such as pembrolizumab and capecitabine are permitted during protocol treatment. All of these treatments are delivered routinely as SOC during conventional radiotherapy.
* Unwilling or unable to participate in all required study evaluations and procedures. Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local patient privacy regulations).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Local recurrences | 3 years
  Local recurrence is defined as histologic evidence of ductal carcinoma in situ or invasive breast cancer in the ipsilateral reconstructed breast or chest wall.
Regional recurrences | 3 years
  Regional recurrence is defined as the cytologic, histologic and/or radiographic evidence of disease in the ipsilateral internal mammary, ipsilateral supraclavicular, ipsilateral infraclavicular and/or ipsilateral axillary nodes or soft tissue of the ipsilateral axilla.

SECONDARY OUTCOMES:
complications | 3 years
  CTCAE toxicities: will evaluate the incidence of any reported acute and late radiotherapy complications using the CTCAE 5.0 grading system when possible.

CONTACTS AND LOCATIONS:
Overall Officials: Aftif Khan, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm